CLINICAL TRIAL: NCT06785506
Title: A Dynamic, Multiple-biomarker Approach Aiming for Individualized Treatment of Heart Failure with Preserved Ejection Fraction (ADAPT-HFpEF)
Brief Title: Multiple-biomarker Approach for Individualized Treatment of Heart Failure with Preserved Ejection Fraction
Acronym: ADAPT-HFpEF
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Ikazia Hospital, Rotterdam (Other); Franciscus Gasthuis & Vlietland (Hospital) (Other); OLVG (Network); Free University Medical Center (Other); Noordwest Ziekenhuisgroep (Other)
Responsible Party: Principal Investigator, Isabella Kardys, Prof. dr., MD PhD, Erasmus Medical Center
Other Study IDs: MEC-2022-0408
Record Dates: First submitted 2024-07-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure with Preserved Ejection Fraction; Heart Failure, Diastolic; Chronic Heart Failure
Keywords: HFpEF; Heart failure; preserved ejection fraction; biomarkers
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (EDTA plasma, citrate plasma, serum) and urine samples are taken at the day of inclusion and at follow-up visits, which will be performed every 6 months, until the end of the scheduled follow-up, or until the patient dies. The maximum total number of samples per patient is 8 (in patients with 3.5 year follow-up).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Heart failure patients visiting the outpatient clinic: Heart failure patients visiting the outpatient clinic

SUMMARY:
The primary objective is to investigate the association between temporal evolutions of blood biomarkers and clinical adverse events, in order to produce a dynamic, individual, and accurate prediction model for patients with HFpEF.

Moreover several secondary objectives will be investigated.

DETAILED DESCRIPTION:
This is a prospective, observational multi-center cohort study which will be conducted at the cardiology departments of the Erasmus Medical Centre (EMC) as well as five other hospitals. A total of 200 HFpEF patients will be included in the study via the outpatient clinics. The follow-up period will constitute a minimum of 2 years and a maximum of 3.5 years. Clinical data will be collected at baseline and blood samples will be collected at baseline and subsequently every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Capable of understanding and signing informed consent
* A diagnosis of HFpEF according to the HFA-PEFF diagnostic algorithm of the ESC or/and a high (90%) probability of HFpEF according to the H2FPEF score, i.e. a score of 6 or higher.

Exclusion Criteria:

* History of LVEF ≤40%
* Scheduled for surgery or intervention for both coronary and non-coronary indication within 6 months of inclusion
* Impaired renal function, defined as eGFR < 20 mL/min/1.73 m2 (CKD-EPI) or requiring dialysis at the time of screening
* Acute or chronic liver disease, defined by serum levels of transaminases or alkaline phosphatase more than three times the upper limit of normal at screening
* COPD Gold stage IV
* Congenital heart disease
* Pregnancy
* Coexistent condition with life expectancy of <1 year
* Unlikely to appear at all scheduled follow-up visits
* Linguistic barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a (suspected) diagnosis of HFpEF will be recruited through the Cardiology outpatient clinics of the Erasmus MC and five other hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the number of participants with a combined endpoint of: urgent visit resulting in intravenous therapy for HF, hospital readmission for acute or worsened HF, and cardiovascular death. | Every 6 months, up to 3,5 years
  This is a composite endpoint; therefore, the first occurrence of any of the described components will result in the endpoint being met for an individual patient.

SECONDARY OUTCOMES:
Number of participants with urgent visit resulting in intravenous therapy for heart failure | Every 6 months, up to 3,5 years
Number of patients with hospital readmission for acute or worsened HF | Every 6 months, up to 3.5 years
Number of participants with cardiovascular death. | Every 6 months, up to 3.5 years
Number of participants with the combined endpoint urgent visit resulting in intravenous therapy for HF, hospital readmission for acute or worsened HF, and all-cause death. | Every 6 months, up to 3,5 years
  This is a composite endpoint; therefore, the first occurrence of any of the described components will result in the endpoint being met for an individual patient.
Number of partcipants with all-cause death | Every 6 months, up to 3,5 years
Number of participants with the combined endpoint of myocardial infarction (fatal and non-fatal), stroke (fatal and non-fatal), percutaneous coronary intervention (PCI) and coronary artery bypass grafting (CABG) | Every 6 months, up to 3,5 years
  This is a composite endpoint; therefore, the first occurrence of any of the described components will result in the endpoint being met for an individual patient.
Number of participants with cardiovascular disease (includes all of the above-mentioned components, except all-cause death) | Every 6 months, up to 3,5 years
  This is a composite endpoint; therefore, the first occurrence of any of the described components will result in the endpoint being met for an individual patient.

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Noordwest Ziekenhuisgroep, Alkmaar, North Holland
  - Amsterdam UMC, Amsterdam, North Holland
  - OLVG Ziekenhuis, Amsterdam, North Holland
  - Franciscus Gasthuis & Vlietland Ziekenhuis, Rotterdam, South Holland
  - Erasmus MC, Rotterdam, South Holland
  - Ikazia Ziekenhuis, Rotterdam, South Holland